CLINICAL TRIAL: NCT00300365
Title: A Randomized, Double Blind, Placebo Controlled Trial of Pioglitazone and Niacin Extended Release in Non-diabetic Patients With Metabolic Syndrome
Brief Title: Pioglitazone vs Placebo in Combination With Niacin Extended Release on Low HDL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Kos Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 803751; Pionir (Other: University of Pennsylvania)
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Metabolic Syndrome
Keywords: HDL cholesterol; Metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Pioglitazone; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pioglitazone and placebo were overencapsulated

ARMS (2):
- Active Pioglitazone + Open-Label Niacin (Experimental): Intervention: Pioglitazone, initially 30mg, then titrated to 45mg + niacin ER 2.0 g/day + aspirin 325 mg/day
  Interventions: Drug: Pioglitazone; Drug: Niacin ER; Drug: Aspirin
- Placebo +Open-Label Niacin (Placebo Comparator): Intervention: Pioglitazone Placebo + 2.0 g/day Open-Label Niacin + 325 mg/day Aspirin
  Interventions: Other: Placebo; Drug: Niacin ER; Drug: Aspirin

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone, initially 30 mg, then titrated to 45 mg/day
  Other Names: Actos
  Arms: Active Pioglitazone + Open-Label Niacin
Other: Placebo — Pioglitazone placebo
  Arms: Placebo +Open-Label Niacin
Drug: Niacin ER — Niacin ER 2.0 g/day
Drug: Aspirin — asprin 325 mg/day

SUMMARY:
We will test our primary hypothesis that combining niacin extended release (niacin-ER), at a daily dosage of up to 2.0 g with pioglitazone, at a daily dosage of 45 mg will result in a 12% greater increase in HDL-C when compared to niacin-ER monotherapy over 12 weeks in non-diabetic patients with the metabolic syndrome (see Table 1).

DETAILED DESCRIPTION:
This is a two-arm, parallel, double-blind randomized prospective clinical trial. The subjects will be asked to provide informed consent, and then undergo screening for enrollment criteria at the first visit (-5 weeks). The subjects who are eligible, and provide informed consent will return for Visit 2 baseline data (-4 weeks), and then begin the unblinded niacin-ER titration. Specifically, subjects will receive a starting dose of niacin-ER of 500 mg per day, which will be increased in 500 mg increments every week up to a dose of 2000 mg per day. Subjects will need to tolerate at least 1500 mg per day of niacin-ER in order to remain in the study and be randomized. Thus subjects who are unable to tolerate the 2000 mg daily dose of niacin-ER will be taken back to 1500 mg per day for one week and then randomized. Subjects who develop prohibitive side effects at doses less than 1500 mg per day will be discontinued from the study. All subjects who are able to take the target dose of niacin-ER will continue that dose of niacin-ER and come to the General Clinical Research Center (GCRC) to be randomized in a 1:1 fashion to either niacin-ER plus pioglitazone or niacin-ER plus matching placebo for 12 weeks. Pioglitazone will be started at 30 mg and then increased to 45 mg at week 6. This entry design is designed to minimize the differences in mean dose of niacin-ER and dropout rate between study groups.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 75
2. HDL-C ≤ 40 mg/dL for Men and HDL-C < 50 mg/dl for Women*
3. At least two of the following criteria (a, b, c, or d) listed below:

   1. Abdominal obesity (waist circumference: men 40 inches and women 35 inches)**
   2. Blood pressure > 130/>85 mmHg in untreated patients OR use of any antihypertensive agent.
   3. Fasting glucose > 100 mg/dL but < 126 mg/dL
   4. Fasting triglycerides > 150 mg/dL

Exclusion Criteria:

1. Diabetes or use of anti-hyperglycemic medication in the last 3 months (subjects with a fasting blood glucose of > 110 mg/dL will have an oral glucose tolerance test (OGTT) to rule out diabetes mellitus).
2. Subjects on statin therapy may be enrolled, but only if they have been on a stable dose for at least 3 months, and are not expected to require titration of statin therapy during the course of the study.
3. Uncontrolled hypertension (defined as systolic bp > 180, diastolic BP > 100).
4. Triglycerides > 400 mg/dL
5. LDL-cholesterol level > 190 mg/dl
6. History of chronic renal insufficiency (serum creatinine >2.0 mg/dl).
7. History of liver disease or abnormal liver function tests (LFTs) (>2x upper limit normal)
8. Hemoglobin < 10 mg/dL
9. History of congestive heart failure (NYHA Class III or IV)
10. Women who are pregnant or lactating
11. History of a non-skin malignancy within the previous 5 years
12. Any major active rheumatologic, pulmonary, or dermatologic disease or other chronic inflammatory condition
13. Surgery in the last 90 days
14. History of HIV positive
15. Active alcohol or drug abuse
16. Active peptic ulcer disease
17. Gout attack within the past 6 months
18. Participation in an investigational drug study within 6 weeks
19. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful study participation
20. Subjects on warfarin may be enrolled, but they will be excluded from the optional adipose biopsy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rick Samaha, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited and participated in the study from December 2005 and July 2007. Subjects were recruited from the University of Pennsylvania and the Philadelphia Veterans Affairs Medical Center.
Pre-assignment Details: 4 weeks prior to randomization, subjects titrated to 2.0 g/day of niacin extended release. Subjects who could not tolerate niacin were excluded from the study.
Groups:
- Pioglitazone Placebo + Open-Label Niacin + Aspirin: Subjects receiving pioglitazone placebo in combination with niacin ER 2.0 g/daily and aspirin 325 mg
- Active Pioglitazone + Open-Label Niacin + Aspirin: Subjects receiving 45 mg/day active pioglitazone in combination with niacin ER 2.0 g/daily and aspirin 325 mg. Subjects received 30mg/day pioglitazone for 6 weeks, followed by 45 mg/day for another 6 weeks
Period: Overall Study
Arm/Group | Pioglitazone Placebo + Open-Label Niacin + Aspirin | Active Pioglitazone + Open-Label Niacin + Aspirin
Started | 38 | 40
Completed | 34 | 38
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Pioglitazone Placebo + Open-Label Niacin + Aspirin: Subjects receiving pioglitazone placebo in combination with niacin ER 2.0 g/daily and 325 mg aspirin
- Active Pioglitazone + Open-Label Niacin + Asprin: Subjects receiving 45 mg/day active pioglitazone in combination with niacin ER 2.0 g/daily and 325 mg aspirin. Subjects received 30mg/day pioglitazone for 6 weeks, followed by 45 mg/day for another 6 weeks
- Total: Total of all reporting groups
Arm/Group | Pioglitazone Placebo + Open-Label Niacin + Aspirin | Active Pioglitazone + Open-Label Niacin + Asprin | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (12.1) | 49.3 (12.2) | 50.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 27 | 30 | 57
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 26 | 26 | 52
  African American | 10 | 10 | 20
  Asian | 0 | 1 | 1
  Hispanic | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Increase in High Density Lipoprotein Cholesterol (HDL-C) at Baseline and 12 Weeks
Description: Mean increase in HDL-C from baseline (week -4) to 12 weeks post randomization in non-diabetic subjects with low HDL-C and metabolic syndrome. After baseline, all subjects titrated niacin extended release (ER) to 2 grams (g) daily over 4 weeks. Subjects were also given 325 mg aspirin to take 30 minutes before the niacin ER. After 4 weeks, half of the subjects added blinded pioglitazone 30mg/day (milligrams/day) for 6 weeks followed by 45 mg/day for 6 weeks; the other half added placebo. HDL-C was was assessed at baseline and 12 weeks post randomization
Time Frame: Baseline, after 12 weeks of pioglitazone vs placebo
Population: All subjects for whom HDL-C measurements were recorded at baseline (week -4) and 12 weeks post randomization to placebo, niacin ER, and aspirin or pioglitazone, niacin ER, and aspirin
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Pioglitazone Placebo + Open-Label Niacin + Aspirin | Active Pioglitazone + Open-Label Niacin + Asprin
Number analyzed (Participants) | 34 | 38
mg/dL
  Baseline HDL-C | 37.4 [36.0 to 38.8] | 36.2 [34.8 to 37.6]
  HDL-C 12 weeks Post Randomization | 40.6 [38.8 to 42.6] | 44.2 [42.2 to 46.2]
Statistical Analysis 1: Comparison: Pioglitazone Placebo + Open-Label Niacin + Aspirin vs Active Pioglitazone + Open-Label Niacin + Asprin; Test type: Superiority; p < 0.0001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from screening (week -4) to completion of study (week 12), for a total of 16 weeks
Arm/Group | Pioglitazone Placebo + Open-Label Niacin + Aspirin | Active Pioglitazone + Open-Label Niacin + Asprin
Serious Adverse Events (participants affected / at risk) | 3/38 | 2/40
Other Adverse Events (participants affected / at risk) | 16/38 | 15/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone Placebo + Open-Label Niacin + Aspirin (N=38) | Active Pioglitazone + Open-Label Niacin + Asprin (N=40)
Hospitalization for Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hospitalization for Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small Intestinal Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Surgery for Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone Placebo + Open-Label Niacin + Aspirin (N=38) | Active Pioglitazone + Open-Label Niacin + Asprin (N=40)
Leg Edema (Blood and lymphatic system disorders) | 6 (6) | 6 (8)
Flushing (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7)
Itching (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No